CLINICAL TRIAL: NCT03503981
Title: Examining Change Mechanisms in Psychotherapy: Relationship Between Specific Ingredients and Common Factors in Promoting Change.
Brief Title: Examining Change Mechanisms in Psychotherapy
Acronym: CAMP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Modum Bad (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Other Study IDs: CAMPFinsrud
Record Dates: First submitted 2018-01-25; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Psychological Disorder; Anxiety Disorders; Depression; Eating Disorder; Post Traumatic Stress Disorder
Keywords: Process-outcome study; Mechanisms of change
MeSH Terms: conditions — Mental Disorders; Anxiety Disorders; Depression; Feeding and Eating Disorders; Stress Disorders, Post-Traumatic | interventions — Psychotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Anxiety unit: Patients have anxiety as a primary diagnose. Receive treatment for anxiety (CBT and MCT).
  Interventions: Other: Psychotherapy
- Eating disorder unit: Patients have eating disorder as primary diagnose. Receive treatment for their eating disorder (CBT and compassion-focused therapy).
  Interventions: Other: Psychotherapy
- Depression unit: Patients have depression as primary disorder. Receive treatment for their depression (Short-term dynamic therapy, existential therapy and relational psychodynamic therapy).
  Interventions: Other: Psychotherapy
- Family unit: One of the members of the family has a psychological disorder. The treatment is focused towards the family and family dynamics.
  Interventions: Other: Psychotherapy
- Trauma unit: Patients have PTSD and relational trauma as primary diagnosis. Receive stabilizing treatment and exposure therapy.
  Interventions: Other: Psychotherapy

INTERVENTIONS:
Other: Psychotherapy — There are different psychotherapy models offered across the units. All patients receive individual treatment and group therapy or psychoeducative groups.

SUMMARY:
This research project seeks to acquire a deeper understanding of the complex influences of common factors and specific ingredients in psychotherapy. By using frequent process-outcome measures, it will address individualized mechanisms of change in psychotherapy by assessing both between and within patient change processes, using a wide spectrum of change indicators.

DETAILED DESCRIPTION:
The study is a naturalistic study conducted by collecting data from in-patient units at Modum Bad (psychiatric hospital). The sample includes different patient groups with a variety of psychological disorders. Further, sample is gathered from units using different treatment approaches (short-term psychodynamic treatment, cognitive-behavioral treatment, metacognitive therapy, compassion-focused therapy, relational psychodynamic therapy, existential therapy and stabilizing trauma-therapy).

The following specific research questions will be explored:

1. The role of common factors:

   1. What are the relative influences of different common factors such as agreement on task and goals, treatment credibility and 'the real relationship', across treatments and diagnoses?
   2. Do some common factor variables stand out regarding ability to explain variance in outcome and across outcomes?
   3. Do measures of common factors have a consistent effect on outcome across treatment models and diagnoses, or does the explanatory value of common factors vary across diagnose and treatment model?
2. The role of specific change mechanisms (affective, cognitive and meta-cognitive):

   1. To what extent do specific change mechanisms predict change in various outcome domains?
   2. Are these specific change mechanisms equally important predictors, or do they vary across treatment or diagnose?
3. Are there interaction effects between common factors and specific factors across treatment models, patient diagnoses and outcome domain?

Self-report data will be collected three times a week on mechanisms of change and symptoms, established by psychotherapy theory and research evidence as important for psychological change. The data collection consists of three different forms administered once per week on different days. The forms are separated by topic; symptoms, contextual factors, and change processes. The questions in the forms are selected from short instruments with good psychometric qualities. The data collection procedure has at present been tested on five patient cohorts with good results.

ELIGIBILITY:
Inclusion Criteria:

* Must be a patient at Modum Bad
* Have a psychological disorder
* Must have rights to treatment according to the rules of specialist health care in Norway. Includes the following:

  1. Patient is expected to have poorer prognosis of life quality if not given treatment
  2. It is expected that the patient will benefit from treatment
  3. It is expected that there is a reasonable cost-effect balance regarding the treatment given and the patient's benefit from treatment.

Exclusion Criteria:

* Acute suicidality
* Ongoing/active abuse of harmful drug(s)
* Under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients accepted for inpatient treatment at Modum Bad Psychiatric hospital during the time of data collection will participate in this study, contingent on consent.
  The patients included will be all genders, adults and reciving treatment from specialist health care.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-08-20 (Estimated); Study Completion 2021-08-20 (Estimated)

PRIMARY OUTCOMES:
Symptom checklist revised (SCL-90-R) | Change measure (baseline, 14 weeks, and 12 months).
  A general measure of symptoms distress

SECONDARY OUTCOMES:
Inventory of interpersonal problems | Change measure (baseline, 14 weeks, and 12 months).
  Self-report questionnaire of interpersonal problems
Beck's depression inventory | Change measure (baseline, 14 weeks, and 12 months).
  Measure of depressive symptoms
PTSD checklist for Diagnostic and Statistical Manual 5 (PCL-5) | Change measure (baseline, 14 weeks, and 12 months).
  PTSD symptom measure
M-POQ outcome, anxiety | Change measure (baseline, 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks, 7 weeks, 8 weeks, 9 weeks, 10 weeks, 11 weeks, 12 weeks, 13 weeks and 14 weeks).
  Measures anxiety symptoms
M-POQ outcome, depression | Change measure (baseline, 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks, 7 weeks, 8 weeks, 9 weeks, 10 weeks, 11 weeks, 12 weeks, 13 weeks and 14 weeks).
  Measures depression symptoms
M-POQ outcome, loneliness | Change measure (baseline, 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks, 7 weeks, 8 weeks, 9 weeks, 10 weeks, 11 weeks, 12 weeks, 13 weeks and 14 weeks).
  Measures experienced loneliness
M-POQ outcome, resilience | Change measure (baseline, 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks, 7 weeks, 8 weeks, 9 weeks, 10 weeks, 11 weeks, 12 weeks, 13 weeks and 14 weeks).
  Measures experienced recilience
M-POQ outcome, well-being | Change measure (baseline, 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks, 7 weeks, 8 weeks, 9 weeks, 10 weeks, 11 weeks, 12 weeks, 13 weeks and 14 weeks).
  Measures experienced well-being

CONTACTS AND LOCATIONS:
Locations (1):
- Modum Bad, Vikersund, Buskerud, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Finsrud I, Nissen-Lie HA, Ulvenes P, Melsom L, Vrabel K, Wampold B. Confidence in the therapist and confidence in the treatment predict symptomatic improvement week by week in therapy: A latent curve modeling approach. J Couns Psychol. 2022 Nov;69(6):823-834. doi: 10.1037/cou0000640. Epub 2022 Sep 22. PMID 36136794
- [Derived] Finsrud I, Nissen-Lie HA, Vrabel K, Hostmaelingen A, Wampold BE, Ulvenes PG. It's the therapist and the treatment: The structure of common therapeutic relationship factors. Psychother Res. 2022 Feb;32(2):139-150. doi: 10.1080/10503307.2021.1916640. Epub 2021 May 2. PMID 33938407